CLINICAL TRIAL: NCT05828225
Title: A Study on the Safety and Efficacy of Chimeric Antigen Receptor T Cells in the Treatment of Refractory Myasthenia Gravis
Brief Title: Evaluate the Safety and Efficacy of CAR-T Cells in the Treatment of Refractory Myasthenia Gravis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2023006
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Myasthenia Gravis
  Interventions: Drug: CD19 CAR-T cells injection

INTERVENTIONS:
Drug: CD19 CAR-T cells injection — CD19 CAR-T in the Treatment of Refractory Myasthenia Gravis

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD19 CAR-T therapy for patients with refractory myasthenia gravis, and to evaluate the pharmacokinetics of CD19 CAR-T in patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 and gender unlimited；
* 2. Confirmed as refractory myasthenia gravis with AchR antibody positive and accord one of the following three conditions

  1. Repeated electrical stimulation suggests neuromuscular conduction deficits；
  2. Tensilon test and neostigmine test positive;
  3. The doctor judged that the symptoms of MG improved after treatment with oral cholinease inhibitors;
* 3. Consistent with the clinical classification of MGFA myasthenia gravis IIa-IVb (including IIa，IIb，IIIa， IIIb， IVa，IVb)
* 4. The baseline MG-ADL score ≥5 and the musculi oculi related score< 50 ；
* 5. Baseline QMG score>11;
* 6. Regular treatment with poor efficacy and/or lack of effective treatment means that there is still recurrence or exacerbation after treatment with conventional hormones, immunosuppressants (such as azathioprine, mycophenolate mofetil, tacrolimus, cyclosporine A, cyclophosphamide, etc.) or rituximab；
* 7. The estimated survival time is more than 12 weeks;
* 8. Women of childbearing age who have negative urine pregnancy test before medication administration and agree to take effective contraceptive measures during the trial period until the last follow-up.

Exclusion Criteria:

* 1. Epilepsy history or other central nervous system disease;
* 2. During the screening visit, the patient's thymectomy was less than 12 months or thymectomy was necessary during the study period or thymic radiation therapy ;
* 3. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythm ia in the past;
* 4. Pregnant (or lactating) women;
* 5. Patients with severe active infections;
* 6. Active infection of hepatitis B virus or hepatitis C virus;
* 7. Systemic steroids have used in the 4 weeks before participating in the treatment (except recently or currently using inhaled steroids);
* 8. Those who have used any gene therapy products before;
* 9. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 10. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0 mg /dl;
* 11. Those who suffer from other uncontrolled diseases are not suitable to join the study;
* 12. HIV infection;
* 13. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD19 CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 90 days after CD19 CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]
Maximum tolerable dose | From date of initial treatment to Day 28 post CD19 CAR-T infusion.
  Maximum tolerable dose

SECONDARY OUTCOMES:
Changes in serum AchR antibody titer | days 7, 14, 21, 28 and 90
  Changes in serum AchR antibody titer
MG-activities of daily living profile (MG-ADL) | Baseline up to 28 days after CD19 CAR T-cells infusion
  MG-ADL Myasthenia Gravis Daily Activity Scale
MG-activities of daily living profile (QMG) | Baseline up to 28 days after CD19 CAR T-cells infusion
  Quantitative Score for Myasthenia Gravis
Myasthenia Gravis Composite Scale (MGC) | Baseline up to 28 days after CD19 CAR T-cells infusion
  Myasthenia Gravis Composite Scale
MG-QOL15 scale | Baseline up to 28 days after CD19 CAR T-cells infusion
  MG-QOL15 Quality of Life Scale for Myasthenia Gravis (15 items)

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China